CLINICAL TRIAL: NCT04721613
Title: Circadian Melatonin Rhythms in Critically Ill Patients With Delirium - A Prospective Single-centre Observational Proof-of-concept Study
Brief Title: Circadian Melatonin Rhythms in Critically Ill Patients With Delirium
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Centre for Chronobiology, Transfaculty Research Platform Molecular and Cognitive Neurosciences (MCN), Psychiatric Hospital of the University of Basel (UPK) (Unknown)
Responsible Party: Sponsor
Other Study IDs: BASEC_01_2021
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: ICU Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hypoactive ICU delirium
  Interventions: Other: Assessment of Melatonin level
- Hyperactive or mixed ICU delirium
  Interventions: Other: Assessment of Melatonin level
- Critically ill patients not suffering form ICU delirium
  Interventions: Other: Assessment of Melatonin level

INTERVENTIONS:
Other: Assessment of Melatonin level — Measuring the plasma or serum melatonin in pg/ml during the first 24 hours after delirium diagnosis in two-hour intervals.

SUMMARY:
Delirious patients often suffer from sleep disturbances such as insomnia, sleep fragmentation, daytime somnolence, and reversal of sleep-wake rhythms. There is evidence, that patients suffering from hyperactive, as well as hypoactive and mixed delirium suffer from disturbed circadian rhythm. The investigators hypothesize that the circadian melatonin profile in critically ill delirious patients measured at two-hourly intervals deviates significantly in terms of phase, width and amplitude from non-delirious critically ill patients with similar age and SOFA (Sequential Organ Failure Assessment) score.

DETAILED DESCRIPTION:
Delirium is a highly prevalent neuropsychological condition in patients admitted to the ICU. Occurrence of a delirium in critically ill patients is associated with prolonged ICU stay and longer hospitalization, reduced quality of life and increased mortality. Furthermore, it is accompanied by a higher risk of cognitive disorder after ICU discharge.

Delirium is defined as an acute, usually reversible state of disturbance of consciousness with a change of perception and cognition. Its fluctuating course leads to a division in three subgroups: hyperactive, hypoactive and mixed delirium. Hyperactive delirious patients present agitated and anxious behaviour, hypoactive delirium however is characterised by withdrawal, somnolence and reduced responsiveness to stimuli. The mixed subtype shows alternating characteristics from both hyperactive and hypoactive delirium.

ICU patients especially in the post-operative setting frequently show several risk factors for delirium, including environmental changes, advanced age, alcohol abuse, dementia, demand for vasopressors, increased doses of opioids or metabolic disturbances.

Sleep and many symptoms that occur in delirium are influenced by the circadian timing system and therefore are thought to be closely related. The neurohormone melatonin plays a major role in regulating circadian rhythms. It is produced in the pineal gland and its diurnal secretion pattern is under the control of the central circadian pacemaker located in the suprachiasmatic nuclei of the anterior hypothalamus. Under normal entrained condition melatonin starts to increase one to three hours prior habitual bedtime, which often coincides with the onset of darkness outside. Thus, melatonin is often referred to as the hormone of darkness. Peak melatonin levels occur approximately two hours prior usual rise time (usually between 2 and 5 A.M.). Melatonin levels are lower during daytime independent of experienced light levels.

Delirious patients often suffer from sleep disturbances such as insomnia, sleep fragmentation, daytime somnolence, and reversal of sleep-wake rhythms. There is evidence that hyperactive as well as hypoactive and mixed delirium is connected to disturbed circadian rhythm. This leads to the question whether there is a link between delirium syndromes as well as different delirium subtypes and potential alterations in circadian melatonin plasma levels compared to non-delirious patients.

Plasma melatonin levels can be assessed in saliva, blood and urine. Due to its rapid metabolisation plasma melatonin levels represent a precise proxy of the current pineal secretion. It therefore is reasonable to collect plasma samples for melatonin assessments frequently throughout the study period to obtain an accurate time course of the circadian melatonin rhythm profile.

There is suggestive evidence that regulating melatonin levels during delirium lowers the incidence of delirium and leads to a reduction of duration and severity of the disorder.

The investigators hypothesize that the circadian melatonin profile in critically ill delirious patients measured in two-hourly intervals across 24 hours deviates significantly from non-delirious critically ill patients with similar age and SOFA (Sequential Organ Failure Assessment) score in terms of phase, width and amplitude.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (aged 55 years or older)
2. Admission to the ICU
3. Current delirium (ICDSC ≥4)
4. Functioning venous or arterial line for blood sample collection

Exclusion Criteria:

1. Delirium prior to ICU admission
2. Intake of beta blockers within 48 hours before study inclusion and during study period
3. Premenopausal women
4. Terminal state
5. Dementia
6. Substance abuse including alcohol in current medical history

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will include 20 patients that fulfil inclusion criteria and do not complete any of the exclusion criteria. Half of the patients should suffer from a hyperactive/mixed delirium with a RASS score ≥2, the other half from a hypoactive delirium. For the control group of 10 patients, the investigators will select age-matched patients grouped in a range of ten years with a minimum of 55 years (55-64 years, 65-74 years, 75-84 years, 85-94 years and higher). The patients of both groups will be hospitalized in the ICU also meeting a similar SOFA score (difference +/- one point). Five patients of the control group will be matched with hyperactively/mixed delirious patients, the other five patients with hypoactively delirious patients.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Melatonin profile | 24 hours
  Difference in melatonin profile in ICU patients with delirium compared to non-delirious patients

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided